CLINICAL TRIAL: NCT04813783
Title: The Effect of Mucositis Care Training Given to Caregivers in Pediatric Leukemia Cases on Mucosal Barrier Damage
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, SEDA ARDAHAN SEVGİLİ, Research Assistant, Ege University
Other Study IDs: 20-6.1T/62
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Leukemia; Mucositis; Nursing Care; Pediatric ALL
MeSH Terms: conditions — Leukemia; Mucositis; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: The first group of 26 volunteers who meet the inclusion criteria of the study will form the control group. These participants will be given clinical routine training about mucositis care.
- Intervention Group: In the study, in order to prevent/minimize the flow of information between the control and intervention groups, the data of the control group will be collected first. Data collection will be suspended in the clinic for three months after the control group data is completed. After this period, data of the enterprise group will be collected. Participants in the intervention group will be provided with mucositis training within the scope of the Mucositis Care Protocol in line with the MASCC / ISOO 2019 Recommendations.
  Interventions: Other: Mucositis care training to be given in line with MASCC / ISOO 2019

INTERVENTIONS:
Other: Mucositis care training to be given in line with MASCC / ISOO 2019 — Mucositis care training to be given in line with MASCC / ISOO 2019
  Groups: Intervention Group

SUMMARY:
There are studies in the literature that include parent training for the prevention and care of mucositis.

Many national and international organizations have emphasized the responsibility of the nurse in patient education and stated it in the relevant laws and regulations.

The regulations focus on the educative role of the nurse for patients. In pediatric oncology clinics where leukaemia treatment and care is provided, the educational role of the nurse is directed towards the child individual and their family, and determining and meeting the educational needs of the whole family is vital in the nursing management of the child with cancer.

In this context, this study aims to examine the effect of mucositis care training to caregivers of pediatric patients aged 2 to 18 years, on the development of mucositis and the clinic's "mucosal barrier damage, laboratory-confirmed bloodstream infections".

DETAILED DESCRIPTION:
Children who are treated for leukaemia are exposed to a wide variety of chemotherapeutic agents and immunosuppressive treatments during the treatment, therefore they are at high risk of complications. Gastrointestinal mucositis is the leading factor affecting the quality of life of the child among the chemotherapy-related complications.

Gastrointestinal mucositis (GM) can be defined as inflammation or ulceration in the gastrointestinal organs due to chemotherapy treatment. Symptoms of GM include abdominal pain, diarrhoea, bleeding, fatigue, malnutrition, dehydration, electrolyte imbalance, and secondary infections. GM can present in two forms as oral and anal mucositis. Both oral and anal all GMs have negative effects on growth and development in children. One of the main issues of the remedial approach in this regard is the provision of qualified mucositis care. There are studies in the literature that include parent training for the prevention and care of mucositis.

Many national and international organizations have emphasized the responsibility of the nurse in patient education and stated it in the relevant laws and regulations. The regulations focus on the educative role of the nurse for patients. In pediatric oncology clinics where leukaemia treatment and care is provided, the educational role of the nurse is directed towards the child individual and their family, and determining and meeting the educational needs of the whole family is vital in the nursing management of the child with cancer.

In this context, this study aims to examine the effect of mucositis care training to caregivers of pediatric patients aged 2 to 18 years, on the development of mucositis and the clinic's "mucosal barrier damage, laboratory-confirmed bloodstream infections".

ELIGIBILITY:
Inclusion Criteria:

* The case is between the ages of 2-18
* The patient is followed up in the Pediatric Hematology Clinic
* The patient is only receiving leukaemia treatment
* The patient is receiving chemotherapy suitable for the high-risk group (T-ALL, High Risk ALL [Protocol HR1-2-3], Middle Risk ALL [Protocol M, Mtx 5gr / m2] The patient does not have any other chronic disease
* The patient does not have a systemic infection
* The patient has a central venous catheter or port catheter Volunteering of the mother and the caregiver parent
* The caring parent knows Turkish and is open to communication

Exclusion Criteria:

-

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of the study will be the cases in the 2-18 age group followed in the Ege University Faculty of Medicine Children's Hospital Pediatric Hematology Clinic and their primary caregiver parents.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Mucositis knowledge scores of caregivers | change from baseline to three days after training
  It is the form prepared by the researchers in line with the literature, questioning the parents' knowledge of the definition of oral/anal mucositis and the application of care principles in mucositis.
change of weight | change from baseline to seven days after training
  change in the child's body weight
change of the degree of mucositis | through study completion, an average of 2 weeks
  the change in the child's mucositis by using WHO Mucositis Scale
change of pain level due to mucositis with WB Scale | through study completion, an average of 2 weeks
  It is the form that includes the pain assessment scale suitable for the child's age. The Wong-Baker Facial Pain Scale will be used for children aged 2 months to 6 years
change of pain level due to mucositis with Numeric Pain Scale | through study completion, an average of 2 weeks
  It is the form that includes the pain assessment scale suitable for the child's age. The Numerical Pain Scale for children aged 7 and above.
Change of Pediatric Oral / Anal Mucositis Care Skills | change from baseline to three days after training
  It is a form prepared by researchers in line with the literature in which the skills of parents regarding the application of care principles in oral / anal mucositis are questioned.
Change of Mucosal barrier injury laboratory-confirmed bloodstream infection rate | change from baseline to seven days after training
  It is a test to eveluate mucosal barrier injury laboratory-confirmed bloodstream infection rate
oral mucositis area measurement | change from baseline to seven days after 21 days
  The measurement will be evaluated with IMITO Wound Application

CONTACTS AND LOCATIONS:
Overall Officials: SELMİN ŞENOL, Study Chair — KÜTAHYA UNIVERSITY
Locations (1):
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No